CLINICAL TRIAL: NCT06929624
Title: A Phase 3, Open-label, Randomized Study of SHR-A1912 Combined With Rituximab + Gemcitabine + Oxaliplatin (R-GEMOX) Versus R-GEMOX in Patients With Relapsed or Refractory Diffuse Large B-cell Lymphoma
Brief Title: A Phase 3 Clinical Study of SHR-A1912 Combined With R-GemOx Versus R-GemOx in Diffuse Large B-cell Lymphoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1912-301
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Gemcitabine; Injections; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-A1912 combined with Rituximab + Gemcitabine + Oxaliplatin (Experimental)
  Interventions: Drug: SHR-A1912 Injection; Drug: Rituximab Injection; Drug: Gemcitabine Hydrochloride for Injection; Drug: Oxaliplatin Injection
- Rituximab + Gemcitabine + Oxaliplatin (Active Comparator)
  Interventions: Drug: Rituximab Injection; Drug: Gemcitabine Hydrochloride for Injection; Drug: Oxaliplatin Injection

INTERVENTIONS:
Drug: SHR-A1912 Injection — SHR-A1912 injection.
  Arms: SHR-A1912 combined with Rituximab + Gemcitabine + Oxaliplatin
Drug: Rituximab Injection — Rituximab injection.
Drug: Gemcitabine Hydrochloride for Injection — Gemcitabine hydrochloride for injection.
Drug: Oxaliplatin Injection — Oxaliplatin injection.

SUMMARY:
This is a multicenter, randomized, open-label, phase 3 clinical study to evaluate the efficacy of SHR-A1912 combined with R-GemOx in relapsed refractory diffuse large B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diffuse large B-cell lymphoma (DLBCL).
2. Have received ≥1 line of systemic antitumor therapy.
3. At least one bi-dimensionally measurable lesion.
4. Expected survival of at least 3 months.
5. Age ≥18 years old and under 80 years old.
6. The patients voluntarily participated in the study, signed informed consent, had good compliance and were willing to cooperate with follow-up.

Exclusion Criteria:

1. Central nervous system lymphoma involvement.
2. Primary mediastinal (thymus) large B-cell lymphoma.
3. Patients who have only one prior line therapy and are candidates for stem cell transplantation.
4. A history of immunodeficiency.
5. A history of severe cardiovascular disease.
6. A history of other malignancies within 5 years prior to administration of the first dose.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Complete response rate (CRR) | Up to 1 years following the first dose of the last enrolled patient.
Overall survival (OS) | Up to 5 years following the first dose of the last enrolled patient.

SECONDARY OUTCOMES:
Adverse events (AEs) | Up to 5 years following the first dose of the last enrolled patient.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided